CLINICAL TRIAL: NCT04561115
Title: A Phase 3, Multicenter, Open-label, Single-sequence, Cross-over, Bioequivalence Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of IVIG-PEG Compared to Gamunex-C in Subjects With Primary Humoral Immunodeficiency
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Immune Globulin (Human) 10% (Gamunex-C) PEG Process (IVIG-PEG) Compared to Gamunex-C in Participants With Primary Humoral Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC1902
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra

STUDY DESIGN:
Intervention Model Description: The study model for this is Single-Sequence crossover.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gamunex-C (Active Comparator): Participants received Gamunex-C by means of an infusion pump at a dose of 200 to 800 mg/kg per infusion at an infusion rate of 1 mg/kg/min or up to 8 mg/kg/min depending on participant tolerance. The participant's usual mg/kg dose (given on either a 3 or 4 week repeating schedule) was the same mg/kg dose and schedule that the participant was receiving prior to entering screening. This mg/kg dose and schedule were used throughout the study duration. Gamunex-C was administered every 3 weeks (±4 days) or 4 weeks (±4 days), depending on the participant's prior IVIG dosing schedule. The duration of Gamunex-C treatment included the Gamunex-C PK Phase (up to 4 weeks) plus the additional Gamunex-C Run-in Phase (up to 4.5 months) for participants not receiving Gamunex-C or not on a stable dose of Gamunex-C upon entering the trial. The approximate maximum duration was up to 6 months.
  Interventions: Biological: Gamunex-C
- IVIG-PEG (Experimental): Participants received IVIG-PEG by means of an infusion pump at a dose of 200 to 800 mg/kg per infusion at an infusion rate of 1 mg/kg/min or up to 8 mg/kg/min depending on participant tolerance. IVIG-PEG was administered every 3 weeks (±4 days) or 4 weeks (±4 days), depending on the participant's prior IVIG dosing schedule. The duration of IVIG-PEG treatment included the IVIG-PEG Treatment Phase (up to 4.5 months) and the IVIG-PEG PK Phase (up to 4 weeks), for an approximate maximum of up to 6 months.
  Interventions: Biological: IVIG-PEG

INTERVENTIONS:
Biological: Gamunex-C — Intravenous infusion.
  Other Names: IVIG-C
  Arms: Gamunex-C
Biological: IVIG-PEG — Intravenous infusion.
  Arms: IVIG-PEG

SUMMARY:
The purpose of this study is to demonstrate bioequivalence of IVIG-PEG with Gamunex-C (IVIG-C) at steady-state as determined by comparing total Immunoglobulin G (IgG) area under the concentration-time curve during the defined dosing interval ([AUC0-τ] either every 3 weeks [AUC0-21 days] or every 4 weeks [AUC0-28 days]) and maximum concentration in a dosing interval (Cmax) in participants diagnosed with primary humoral immunodeficiency (PI) currently receiving chronic IVIG replacement treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age (inclusive) at Screening
* Documented and confirmed pre-existing diagnosis of PI with features of hypogammaglobulinemia requiring IV IgG replacement therapy including but not limited to the following humoral-based immunodeficiency syndromes (example, X-linked agammaglobulinemia, common variable immunodeficiency), and combined immunodeficiency syndromes without lymphocytopenia (example, hyper immunoglobulin M [IgM] immunodeficiency syndrome).
* IgG trough level ≥500 milligrams per deciliter (mg/dL) at screening visit. Note: Patients entering Group 1 must additionally have trough levels ≥500 mg/dL documented within the previous year. For patients entering Group 2, if Screening trough levels are not ≥500 mg/dL, the subject will be a Screen Failure, but may be rescreened following dose adjustment of their original IV IgG replacement therapy regimen and recording an IgG trough level ≥500 mg/dL
* Has not had an SBI within the last 6 months prior to screening or during the screening.
* Medical records are available to document diagnosis, previous infections, and treatment.
* Willing to comply with all aspects of the study protocol, including blood sampling, for the duration of the study.
* Signed and dated a written informed consent form (ICF) confirming his or her willingness to participate in study GC1902.

Exclusion Criteria:

* Has an acquired medical condition that is known to cause secondary immune deficiency such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000per microliters (1000/μL) [1.0 x 10^9/L]), or human immunodeficiency virus (HIV) infection/acquired immune deficiency syndrome (AIDS).
* Has known selective Immunoglobulin A (IgA) deficiency (with or without antibodies to IgA). (Note: exclusion is for the specific diagnostic entity. It does not exclude other forms of primary humoral immunodeficiency which have decreased IgA in addition to decreased IgG requiring IgG replacement).
* Has isolated IgG subclass deficiency or an isolated specific antibody deficiency disorder, or transient hypogammaglobulinemia of infancy
* The subject has had a known serious adverse reaction to immunoglobulin or any severe anaphylactic reaction to blood or any blood-derived product.
* Has a history of thrombotic complications following IVIG therapy.
* Has a history of or current diagnosis of deep venous thrombosis (DVT) or thromboembolism (e.g., myocardial infarction, cerebrovascular accident or transient ischemic attack); history refers to an incident in the year prior to the Screening Visit or 2 episodes over lifetime or has thrombosis risk factors (e.g., prolonged immobilization, use of estrogens, indwelling central vascular catheters).
* Has a known hyperviscosity syndrome or hypercoagulable states.
* Has liver enzyme levels (alanine aminotransferase [ALT], aspartate aminotransferase [AST], gammaglutamyl transferase [GGT], or lactate dehydrogenase [LDH]) greater than 2.5 times the upper limit of normal (ULN) at the screening visit as defined by the testing laboratory.
* Has pre-existing renal impairment (defined by serum creatinine greater than 1.5 times the ULN or blood urea nitrogen [BUN] greater than 2.5 times the ULN, or any subject who is on dialysis) at the screening visit or any history of acute renal injury.
* Has clinically significant history of drug or alcohol abuse or dependence in the opinion of the Investigator (must be within the past 12 months and noted in the subject's medical records or documented at screening).
* Clinical evidence of any significant acute or chronic medical condition (e.g., renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing state) that, in the opinion of the Investigator, may interfere with the conduct of the study or may place the subject at undue medical risk.
* Females of childbearing potential who are pregnant, have a positive pregnancy test at Screening (human chorionic gonadotropin [HCG]-based assay), are breastfeeding, or unwilling to practice a highly effective method of contraception (eg, oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device [IUD] or intrauterine system [IUS], condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study. Note: True abstinence: When this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception).
* Receiving any of the following medications: (a) immunosuppressants including chemotherapeutic agents, (b) immunomodulators, (c) long-term systemic corticosteroids defined as daily dose >1 mg of prednisone equivalent/kg/day for >30 days. Note: Intermittent courses not exceeding >1mg of prednisone equivalent/kg/day for >30 days would not exclude the subject. Inhaled or topical corticosteroids are allowed.
* Has uncontrolled arterial hypertension (systolic blood pressure [SBP] >160 mm Hg and/or diastolic blood pressure [DBP] >100 mm Hg)
* Has hemoglobin <11 g/dL at the Screening Visit
* Unable or unwilling to provide a storage serum sample at the Screening Visit. Note: A pre-treatment serum sample to be stored at -94°F (-70ºC) for possible future testing is required.
* Received any live virus vaccine within 5 months prior to the Screening Visit and not willing to postpone receiving any live virus vaccines until 6 months after completing study treatment
* Has a known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has participated in another clinical trial within 30 days prior to Screening or has received any investigational product, with the exception of other IgG products, within the previous 3 months prior to the Screening Visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Alabama Allergy & Asthma Center, Birmingham, Alabama
  - Allergy Associates of the Palm Beaches PA, North Palm Beach, Florida
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Washington University, St Louis, Missouri
  - Optimed Research, LLC, Columbus, Ohio
  - Allergy, Asthma and Immunology Center, P.C., Tulsa, Oklahoma
  - Allergy Partners of North Texas Research, Dallas, Texas
  - AARA Research Center, Dallas, Texas
  - Allergy, Asthma & Immunology Clinic, P.A., Irving, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 investigative sites in the United States from 02 September 2020 (first participant enrolled to receive the study drug) to 28 March 2022 (last participant completed).
Pre-assignment Details: A total of 43 participants were screened, of which 33 participants received study treatment. 22 participants entered the Gamunex-C (GC) Run-in Phase and received GC treatment to achieve an approximate steady-state condition prior to entering the GC pharmacokinetic (PK) Phase as per investigators discretion. Eleven (11) participants directly entered into the GC PK phase.
Groups:
- Gamunex-C: Participants received GC by means of an infusion pump at a dose of 200 to 800 mg/kg per infusion at an infusion rate of 1 mg/kg/min or up to 8 mg/kg/min depending on participant tolerance. The participant's usual mg/kg dose (given on either a 3 or 4 week repeating schedule) was the same mg/kg dose and schedule that the participant was receiving prior to entering screening. This mg/kg dose and schedule were used throughout the study duration. GC was administered every 3 weeks (±4 days) or 4 weeks (±4 days), depending on the participant's prior IVIG dosing schedule. The duration of GC treatment included the GC PK Phase (up to 4 weeks) plus the additional GC Run-in Phase (up to 4.5 months) for participants not receiving GC or not on a stable dose of GC upon entering the trial. The approximate maximum duration was up to 6 months.
Period: GC Run-in Phase (Up to 4.5 Months)
Arm/Group | Gamunex-C | IVIG-PEG
Started | 22 (Participants not on stable GC treatment entered the GC Run-in Phase to receive GC treatment to achieve an approximate steady-state condition prior to entering the GC PK Phase.) | 0
Completed | 22 | 0
Not Completed | 0 | 0
Period: GC Run-In + PK Phase (Up to 6 Months)
Arm/Group | Gamunex-C | IVIG-PEG
Started | 33 (11 participants directly entered GC PK Phase.) | 0
Completed | 32 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: IVIG-PEG Treatment (Up to 4.5 Months)
Arm/Group | Gamunex-C | IVIG-PEG
Started | 0 | 32
Completed | 0 | 31
Not Completed | 0 | 1
Not completed — The Dose Changed Back and Forth 800-600 Mg/Kg During GC Phase Fulfilling Discontinuation Criteria | 0 | 1
Period: IVIG-PEG + PK Phase (Up to 6 Months)
Arm/Group | Gamunex-C | IVIG-PEG
Started | 0 | 32
Completed | 0 | 31
Not Completed | 0 | 1
Not completed — The Dose Changed Back and Forth 800-600 Mg/Kg During GC Phase Fulfilling Discontinuation Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or Gamunex-C).
Arm/Group | Gamunex-C
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-7): Area Under the Concentration Time Curve Over a Dosing Interval of Either Every 3 Weeks [AUC0-21 Days] or Every 4 Weeks [AUC0-28 Days] for Total Immunoglobulin G (IgG)
Description: AUC (0-7 days) is calculated as AUC (0-21 days)/3 for subjects with a dosing frequency of every 3 weeks and as AUC(0-28 days)/4 for subjects with a dosing frequency of every 4 weeks.
Time Frame: Pre-dose, within 10 minutes of last infusion completion, at 1, 3, 6, 24, 48 hours and 4, 7, 14 and 21 days (up to 3 weeks), and 28 days (up to 4 weeks - only for subjects on a 4-week dosing schedule) post-infusion
Population: The PK population consisted of all participants who received study drug and had sufficient and valid total IgG concentration versus time data for either the IVIG-PEG PK Phase or GC PK Phase to allow calculation of AUC0-τ. Overall number analyzed are the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: hour*milligrams per decilitres (h*mg/dL)
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 29 | 31
hour*milligrams per decilitres (h*mg/dL) | 232088.8 (32848.46) | 219149.9 (36894.29)
Statistical Analysis 1: Comparison: Gamunex-C vs IVIG-PEG; Test type: Equivalence — The relative alpha level for statistical significance was 0.1 (alpha=0.05 for one-sided test), or a 90% CI was used for the bioequivalence test; Geometric Least Square Mean Ratio = 0.948, 90% CI 2-sided [0.926 to 0.972]

2. Primary Outcome: Cmax: Maximum Concentration in a Dosing Interval for Total IgG
Time Frame: Pre-dose, within 10 minutes of last infusion completion, at 1, 3, 6, 24, 48 hours, and 4, 7, 14, 21 and 28 days post-infusion (up to 4 weeks)
Population: The PK population consisted of all participants who received study drug and had sufficient and valid total IgG concentration versus time data for either the IVIG-PEG PK Phase or GC PK Phase to allow calculation of AUC0-τ.
Measure: Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 32 | 31
milligrams per decilitre (mg/dL) | 2328.8 (426.73) | 2330.4 (660.99)
Statistical Analysis 1: Comparison: Gamunex-C vs IVIG-PEG; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Least Square Mean Ratio = 0.978, 90% CI 2-sided [0.937 to 1.021]

3. Secondary Outcome: Rate of Serious Bacterial Infections (SBIs)
Description: The rate of SBI events per participant per year during treatment was calculated as the total number of SBI events divided by the total duration of exposure in years across all participants. The 2-sided 98% confidence interval (CI) was determined from a generalized linear model for Poisson regression for the log-transformed number of events with log-transformed duration of exposure in years as an offset variable.
Time Frame: Baseline up to 6 months for each period, i.e., overall GC treatment phase and overall IVIG-PEG treatment phase with an aggregate duration of up to 12 months
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or GC).
Measure: Number (98% Confidence Interval); unit: rate of events per participant per year
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 33 | 32
rate of events per participant per year | 0 [NA to NA] — Here NA signifies that 98% CI was not estimable due to zero number of events. | 0 [NA to NA] — Here NA signifies that 98% CI was not estimable due to zero number of events.

4. Secondary Outcome: Rate of Events Per Participant Per Year in Participants With Any Kind of Infection
Description: Rate of events per participant per year is calculated as the total number of events divided by the total duration of exposure in years across all participants. Any kind of infections included serious/nonserious including acute sinusitis, exacerbation of chronic sinusitis, acute otitis media, pneumonia, acute bronchitis, infectious diarrhea etc.) as determined by the Investigator.
Time Frame: as for outcome 3
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or Gamunex-C).
Measure: Number (95% Confidence Interval); unit: rate of events per participant per year
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 33 | 32
rate of events per participant per year | 1.332 [0.789 to 2.249] | 1.580 [1.041 to 2.400]

5. Secondary Outcome: Rate of Days Per Person Per Year That Participants Were on Antibiotics
Description: Rate of days per person per year is calculated as the total number of days divided by the total duration of exposure in years across all participants. Antibiotics included prophylactic and therapeutic.
Time Frame: as for outcome 3
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or GC).
Measure: Number (95% Confidence Interval); unit: rate of days per participant per year
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 33 | 32
rate of days per participant per year
  Prophylactic Antibiotics | 0 [0.0 to 0.0] | 9.410 [7.929 to 11.167]
  Therapeutic Antibiotics | 28.257 [25.220 to 31.661] | 27.079 [24.479 to 29.956]

6. Secondary Outcome: Number of Participants Hospitalized Due to Infection
Description: Hospitalization was considered only in cases of hospital admission (including emergency room stay) for equal or more than 24 hours.
Time Frame: as for outcome 3
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or GC).
Measure: Count of Participants; unit: Participants
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

7. Secondary Outcome: Rate of Days of Work/School/Daily Activities Missed Per Participant Due to Infections and Their Treatment
Description: Rate of days per person per year is calculated as the total number of days divided by the total duration of exposure in years across all participants.
Time Frame: as for outcome 3
Population: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or GC).
Measure: Number (95% Confidence Interval); unit: rate of days missed/participant per year
Arm/Group | Gamunex-C | IVIG-PEG
Number analyzed (Participants) | 33 | 32
rate of days missed/participant per year | 7.421 [5.944 to 9.265] | 6.177 [5.000 to 7.631]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (Up to Week 54)
Description: The safety population included all participants who received any amount of study drug (IVIG-PEG and/or GC).
Arm/Group | Gamunex-C | IVIG-PEG
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/32
Other Adverse Events (participants affected / at risk) | 20/33 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gamunex-C (N=33) | IVIG-PEG (N=32)
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gamunex-C (N=33) | IVIG-PEG (N=32)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Methylenetetrahydrofolate Reductase Gene Mutation (Congenital, familial and genetic disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Chorioretinal disorder (Eye disorders) | 1 | 0
Eye Inflammation (Eye disorders) | 0 | 1
Eye Pruritus (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Administration site bruise (General disorders) | 1 | 0
Application site rash (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 0
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 0 | 1
Multiple allergies (Immune system disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 2 | 4
Diverticulitis (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1
Helicobacter Gastritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hyphaema (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Traumatic iritis (Injury, poisoning and procedural complications) | 0 | 1
Free Prostate-specific Antigen Increased (Investigations) | 1 | 0
Low Density Lipoprotein Increased (Investigations) | 0 | 1
SARS-CoV-2 Test Positive (Investigations) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Hypoferritinaemia (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 5 | 5
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04561115/Prot_002.pdf
  • Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04561115/SAP_001.pdf